CLINICAL TRIAL: NCT00191399
Title: Bipolar Depression Assessment Study on Tx Response
Brief Title: Bipolar Depression Study: Bipolar Depression Assessment Study on Treatment Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9370; F1D-SU-HGMA
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Depression, Bipolar
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Fluoxetine

INTERVENTIONS:
Drug: Olanzapine
Drug: Fluoxetine

SUMMARY:
The primary objective of this study is to assess the efficacy of olanzapine and fluoxetine combined on all the visits as compared with the baseline visit in patients with bipolar disorder, measured by the total score of the Montgomery-Asberg Depression Rating Scale (MADRS).

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for bipolar depression, in the opinion of the investigator, according to the Diagnostic and Statistical Manual of Mental Disorders [Text Revision] (DSM-IV-TR) disease diagnostic criteria.
* Patients must have experienced, in the opinion of the investigator, at least one previous hypomanic, manic or mixed episode as defined in DSM-IV-TR.
* Subjects must have an initial score at Visit 1 of at least 20 on the MADRS.

Exclusion Criteria:

* Any patient currently meeting DSM-IV-TR criteria rapid-cycling course.
* A CGI-Severity - Mania score of at least 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-05; Study Completion 2006-03

PRIMARY OUTCOMES:
MADRS is a rating scale for severity of depressive mood symptoms.

SECONDARY OUTCOMES:
Clinical Global Impression - Bipolar Version (CGI-BP) Severity - Depression is used by the clinician to record the severity of depression illness at the time of assessment
CGI-BP Severity - Mania is used by the clinician to record the severity of mania illness at the time of assessment
Short Form-12 (SF-12) Questionnaire was developed from the SF-36 Health Survey for use in monitoring outcomes for general and specific populations.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (10):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington, United States
- Puerto Rico (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Caguas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Canovanas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Manatí
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Mayagüez
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Rio Piedras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Santurce

REFERENCES:
- [Derived] Tamayo JM, Sutton VK, Mattei MA, Diaz B, Jamal HH, Vieta E, Zarate CA Jr, Fumero I, Tohen M. Effectiveness and safety of the combination of fluoxetine and olanzapine in outpatients with bipolar depression: an open-label, randomized, flexible-dose study in Puerto Rico. J Clin Psychopharmacol. 2009 Aug;29(4):358-61. doi: 10.1097/JCP.0b013e3181ad223f. PMID 19593175